## Participant Informed Consent for Clinical Research

## Study title for participants: Physician Use of Non-English Language Skills in Cancer Care

Official study title internet search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:

Physician use of Non-English Language Skills in Cancer Care

Subtitle: Patient consent form

Lead Researcher: Lisa Diamond, MD, MPH, 646-888-8061

If you are the parent or legal guardian of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to your child, if the participant is a minor, or to a person with a cognitive impairment for whom you are the Legally Authorized Representative (LAR).

#### **Overview and Key Information**

#### Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

You are being asked to take part in this research study because you have an initial consult meeting between you and your treating cancer doctor. The researchers would like to test a method for analyzing interactions between patients and doctors, the Roter Interaction Analysis System (RIAS). The RIAS measures the quality of communication between patients and their cancer doctors.

#### Taking part in this study is your choice.

You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered.

## What are my other choices if I decide not to take part in this study?

· You may choose to take part in a different research study, if one is available

## What will happen if I decide to take part in this study?

If you decide to take part in the study, we will audio record the initial consult meeting between you and your treating cancer doctor. The audio recording of this session will then be uploaded to a computer and analyzed using the Rother Interaction Analysis System (RIAS). Once analyzed, the audio recording will be destroyed from our study files.

You will be in the study for one day only.



#### What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### Risks

We want to make sure that you know about a few key risks right now. We will also give you more information in the What risks can I expect from taking part in this study? section of this consent form.

If you choose to take part in this study, there is a risk that knowing you are being audio recorded may cause you to become anxious or upset.

There may be some risks that the study doctors do not yet know about.

#### Benefits

Because this study does not provide treatment, you will not receive any health benefit from participating in the study. What we learn from the study may help other people in the future.

#### If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

If you decide you no longer want to be audio recorded during the discussion with your doctor, tell the doctor that you no longer would like to be recorded. The doctor will stop recording the session and you will be taken off the study. Audio recorded information previously recorded will be retained for the study analysis. If you decide to stop participation and prefer not to have any of your appointment discussion kept for research, please let the study staff know and the recording will be destroyed.

#### Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest
- You do not follow the study rules
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or the study sponsor, Memorial Sloan Kettering Cancer Center. The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of



this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

#### What is the purpose of this study?

This study will test a method for analyzing interactions between patients and doctors, the Roter Interaction Analysis System (RIAS). The RIAS measures the quality of communication between patients and their cancer doctors. Clear communication between patients and members of their treating team is an important part of cancer care. For example, understanding your cancer diagnoses, treatment options, and being able to talk freely with your doctor about any concerns are very important parts of cancer care. Communication can be challenging for both English and non-English speaking patients. For non-English speaking patients, although interpreter services are provided free of charge, it can still be difficult to have clear communication with doctors. Being able to measure the quality of communication between clinical providers and patients will be helpful in learning about the problems cancer patients face, and help investigators find a way to address these problems.

There will be about 48 patients taking part in this study and we anticipate about 38 different physicians to participate. Of the 48 patients, about 12 will be from Lincoln Hospital, about 12 will be from Elmhurst Medical Center, about 12 will be from Queens Cancer Center, about 6 will be from Memorial Sloan Kettering Cancer Center, and about 6 will be from Ralph Lauren Center for Cancer Care.

#### What are the study groups?

Study patients will be grouped in pairs with their treating doctor based upon the expected types of communication.

- Group 1 will be Spanish-speaking patients and Spanish-speaking doctors, nurse practitioners, or physician assistants communicating in Spanish
- Group 2 will be English-speaking patients and English-speaking doctors, nurse practitioners, or physician assistants communicating in English
- Group 3 will be Spanish-speaking patients and somewhat fluent Spanish-speaking doctors, nurse practitioners, or physician assistants communicating in Spanish
- Group 4 will be Spanish-speaking patients and English-speaking doctors, nurse practitioners, or physician assistants communicating through an interpreter

## What extra tests and procedures will I have if I take part in this study?

#### Before you begin the main part of the study:

- We will check your medical records to see if you qualify to participate.
- We will also check with your treating doctor to see if you can participate in this study.

#### During the study:

- We will audio record the initial consult meeting between you and your treating cancer doctor.
- The audio recording of this session will then be uploaded to a computer and analyzed using the Roter Interaction Analysis System (RIAS).
- Once analyzed, the audio recording will be destroyed from our study files.

There are no extra tests or procedures asked of you if you take part in this study.

#### Will I receive the results of my research tests?



IRB Number: 15-316 A(15) Approval date: 03-Oct-2019

Neither you nor your doctor will receive the results of any tests done for research purposes during this study.

## What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office.
- You may be asked sensitive or private questions that you do not usually discuss.
- · Knowing you are being audio recorded may cause you to become anxious or upset.
- During the session, tell your doctor if at any time you feel uncomfortable and would like to stop audio recording.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor does not know who will or will not have side effects.

Let the study doctor know of any questions you have about any concerns you may have.

#### What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments
- Tell the study doctor about:
  - All medications and any supplements you are taking
  - Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - Whether you have been or are currently in another research study
- Let the study doctor know if you skipped or chose not to answer any of the questions in the questionnaire/survey.

#### Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Center.

The study is funded by National Institutes of Health.

No conflicts of interest have been identified for either the institution or the investigator(s) in this study.

## What are the costs of taking part in this study?

There is no cost for taking part in this study. We are asking to audio record and analyze the initial clinical appointment between you and your treating doctor at no charge to you.

#### Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.



#### Memorial Sloan Kettering Cancer Center IRB Number: 15-316 A(15) Approval date: 03-Oct-2019

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company.

If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.

#### Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.

In the future, your information (data) may be de-identified, which means that your data will be assigned a unique code, and the list that links the code to your name will be stored separately from your data. Your de-identified information may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK, and may be stored in public databases. All requests for data sharing will be reviewed by the study sponsor, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or social security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.

Some of your health information from this study will be kept in a central database for research. Your name and contact information will be stored in the database.

The study doctors have a Certificate of Confidentiality from the National Institutes of Health for this study. This gives MSK an additional way to protect sensitive information that identifies you in your records if it is requested as part of a legal proceeding. However, MSK may still be required to share some of your medical information if required by law.



Memorial Sloan Kettering Cancer Center IRB Number: 15-316 A(15) Approval date: 03-Oct-2019

#### Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.



#### Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

Physician Use of Non-English Language Skills in Cancer Care

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

# 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

#### 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigator(s): Lisa Diamond, MD, MPH and Francesca Gany, MD, MS
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



Approval date: 03-Oct-2019

#### 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- The company or organization that provides the funding for the study, National Institutes of Health.
- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study procedure.
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)
- Other qualified researchers, approved by Memorial Sloan Kettering Cancer Center, who may receive individual research results that do not identify you.

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

#### 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

#### 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the



# Memorial Sloan Kettering Cancer Center IRB Number: 15-316 A(15) Approval date: 03-Oct-2019

study may be analyzed for many years, and it is not possible to know when this analysis will be completed.

## 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be
  able to participate in this research study. However, if you do not sign, it will not affect your
  ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to your medical record at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

#### Notice concerning HIV-related information

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your rights.



Memorial Sloan Kettering Cancer Center IRB Number: 15-316 A(15) Approval date: 03-Oct-2019

#### Participant Informed Consent/Research Authorization for Clinical Research

#### Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information, including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

| Consenting professional must personally sign and date | | | | |
|---|---|---|---|---|
| Consenting professional's | | | | Date: |
| signature | | | | |
| Consenting professions | ıl's name | | | |
| (Print) | | | | |
| Participant's (or Legally A I have read this form that desc with the consenting profession this clinical research study; (2) information (data about myself of this consent form. | ribes the clini<br>al. By signing<br>to authorize<br>/the participa | ical research study. g below, I agree to the the use and disclos nt); and (3) to state | I have also talked in the following: (1) to ure of my/the partice that I have received | it over to my satisfaction<br>voluntarily participate in<br>cipant's protected health<br>d a signed and dated copy |
| | icipant/L/ | AR must persona | , | |
| Participant/LAR | | | Dat | te: |
| signature | | | | |
| Participant/LAR | | | | |
| name (Print) | | | | |
| LAR relationship to | | | | |
| participant | | | | |
| Witness signature (if recomparticipant's (or LAR's) land for the participant (or LAR) ☐ Other: I confirm that the control of this study by signing this for the participant (or LAR) | peaking partic<br>guage, and I<br>onsent discus | confirm that the corsion occurred, and t | nsent discussion was<br>that the participant | as appropriately interpreted |
| Name of witness: | | | | |
| Signature of witness: (The name of the witness must be documented in the EMR.) | | | | Date: |
| Interpreter (if required) | | | | |
| Name of interpreter (if ) | | | | |
| ID number (if phone int | | | | |
| (The interpreter's name or ID r | | | he EMR.) | |

The participant/Legally Authorized Representative must be provided with a signed copy of this form.

